CLINICAL TRIAL: NCT04460482
Title: Near-infrared Spectroscopy Guided Percutaneous Coronary Intervention in Patients With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Manijeh Noori, MD; PhD-student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: s-20200010
Record Dates: First submitted 2020-07-02; First posted 2020-07-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Myocardial Infarction; Coronary Artery Disease; Myocardial Ischemia; Atherosclerosis; Lipid-Rich Atherosclerosis of Coronary Artery; Vascular Diseases; Infarct Ischemia
Keywords: drug-eluting stent; near-infrared spectrocopy; intravascular ultrasound; optical coherence tomography
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Myocardial Ischemia; Atherosclerosis; Vascular Diseases | interventions — Spectroscopy, Near-Infrared; Angiography

STUDY DESIGN:
Intervention Model Description: Eligible patients randomized to NIRS-guided or standard angiographic-guided intervention with DES
Who Masked: Investigator, Outcomes Assessor
Masking Description: Offline data analyzis are being performed without knowing which intervention group the patients are from
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIRS-guided PCI (Active Comparator): Near-infrared Spectroscopy guided Percutaneous coronary intervention with implantation of drug-eluting stent
  Interventions: Device: Near-infrared spectroscopy (NIRS)
- Angiography-guided PCI (Active Comparator): Angiography-guided percutaneous coronary intervention with implantation of a drug-eluting stent
  Interventions: Device: Angiography

INTERVENTIONS:
Device: Near-infrared spectroscopy (NIRS) — NIRS-guided PCI
  Arms: NIRS-guided PCI
Device: Angiography — Angiography guided PCI
  Arms: Angiography-guided PCI

SUMMARY:
The aim of this study is to investigate whether near-infrared guided percutaneous coronary intervention in patients with acute myocardial infarction provides improved stent strut coverage at six months compared to conventionally angiography guided percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background Myocardial infarction (MI) secondary to atherosclerotic coronary artery disease is mainly due to plaque-rupture with formation of a luminal thrombogenic material. Lesions responsible for MI are more frequently composed of lipid-rich plaques (LRP) in both culprit and in non-culprit lesions compared to lesions in patients with stable angina.

LRP is thought to be main precursor for future coronary events and may also have an impact on complications following percutaneous coronary intervention (PCI). It has been previously indicated that stent thrombosis (ST) and restenosis often occur when stenting a lipid-rich plaque. And if using angiography guidance only during PCI, there is a potential risk of implantation of a stent edge on a lipid pool, which can result in incomplete stent coverage of a lesion. The incidence of restenosis and ST may be related to the lesion characteristics, clinical presentation, antithrombotic treatment and stent design. Other factors may include inflammatory reaction to the polymer coating containing drug that delays vascular healing, insufficient stent strut coverage and incomplete stent apposition (ISA).

Invasive imaging modality can contribute to better understanding of the changes that occur in the vessel wall during stent implantation.

Intravascular ultrasound (IVUS) combined with a new imaging modality called near-infrared spectroscopy (NIRS) can identify LRP and provide a semi-quantitative estimate of amount of LRP present within selected region of interest. The method is excellent to identify ISA and improve stent implantation technique.

Optical coherence tomography (OCT) is a high resolution imaging modality that can analyze healing pattern after stent implantation such as stent strut coverage.

Method The study is designed as a prospective randomized trial conducted at a single center (Odense University Hospital). Patients with MI will be enrolled if they fulfill the criteria. The study is submitted and approved by The Regional Committees on Health Research Ethics for Southern Denmark (Project-ID: S-20200010) and Danish Data Agency (Journal nr.: 20/18008).

Eligible patients will be randomly assigned to either NIRS-guided PCI or conventual angiography-guided PCI with implantation of Everolimus-eluting Xience stent, which is CE marked. NIRS will be performed in both groups after predilation and stent implantation. In NIRS-guided group the analyses will be used to identify LRP, and to measure vessel wall diameter in reference segments and lesion length. In angiography-guided group the analyses will not be available for the PCI operator and are for observation purpose only. OCT will be performed in both groups after stent implantation, but will be only available for interpretation in NIRS-guided group. In case of reintervention in NIRS-guided group, a final OCT will be performed.

Optimal PCI criteria were following: 1) minimum stent area (MSA) ≥ 5.5 mm2 and ≥ 90% of the distal reference lumen area; 2) no major stent malapposition; 3) plaque burden < 50% at stent edge border; 4) LCBI4mm < 150 in reference segments; and 5) no major stent edge dissection. In case of 1-3, we recommended additional post-dilatation, and in case of 4-5 we recommended an additional stent.

A significant LRP was with lipid-core burden index (maxLCBI4mm) ≥ 150.

Patients will be contacted by telephone to evaluate the clinical situation and to reduce the potential risk of dropout. After 6 months OCT will be performed in both groups to evaluate stent strut coverage and vessel healing.

Statistics Assuming data are normally distributed, categorical data will be presented as numbers and frequencies and compared using chi2-test. Continuous data will be presented as mean ± SD and compared using Student t test. SPSS version 26.0 will be used for the statistical analysis.

Sample size calculation Based on a previous study IVUS-guided PCI in STEMI, the percentage of covered stent struts was 85.4%±7.9. We hypothesized that the coverage in angiography-guided group will be lower by 5.6% at 6 month. A sample size of 86 patients (43 patients in each group) was required for the study to have a power of 80% and two-tailed significance level of 0.05. We expected a dropout rate of 20%, and 104 patients were required to be recruited in the trial.

Sato N, Minami Y, Shimohama T, Kameda R, Tojo T, Ako J. Vascular response and intrastent thrombus in the early phase after drug-eluting versus bare-metal stent implantation in patients with ST-segment elevation myocardial infarction: An observational, single-center study. Health Sci Rep. 2019;2(1):e105.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome (ST-elevation myocardial infarction and non-ST elevation myocardial infarction) referred for invasive coronary angiography and percutaneous coronary intervention at Department of Cardiology, Odense University Hospital (Odense, Denmark)

Exclusion Criteria:

* participation in other randomized clinical trials
* life expectancy < 1 year
* allergy to aspirin, clopidogrel, ticagrelor or prasugrel
* eGFR < 30 mL/min
* tortuous and angiographically estimated extremely calcified lesions
* ostial, left main and bifurcation lesions
* lesions in a reference vessel diameter < 2.0 mm
* hemodynamic instability
* Scheduled for coronary artery bypass grafting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Proportion of stent strut coverage | 6 months after index percutaneous coronary intervention
  Proportion of stent strut coverage at 6 months follow up estimated by OCT

SECONDARY OUTCOMES:
Uncovered stent struts | 6 months after index percutaneous coronary intervention
Persistent stent malapposition | 6 months after index percutaneous coronary intervention
Maximal neointimal growth | 6 months after index percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lisette Okkels Jensen, MD PhD Prof, Study Chair — Odense University Hospital
Locations (1):
- Manijeh Noori, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No